CLINICAL TRIAL: NCT03157544
Title: Complementary Management of Chronic Neck and/or Low Back Pain With a Multimodal Non-pharmacological Pain Relief Kit
Brief Title: Complementary Management of Chronic Neck and/or Low Back Pain With a Pain Relief Kit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSR_Toolkit
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Pain, Chronic; Musculoskeletal Pain; Low Back Pain; Neck Pain
Keywords: Chronic Neck Pain; Chronic Back Pain; non-pharmacological; pain relief
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Low Back Pain; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Relief Kit (Experimental): Immediately following baseline data collection participants will be given the Pain Relief Kit and instructed about the contents. From this kit, a sample of Biofreeze® and TheraBand® Kinesiology Tape will be applied to the participant. The contents of the Pain Relief Kit will include four modes of non-pharmacological interventions that have been previously demonstrated to relieve musculoskeletal pain. Following Baseline data collection, participants will review the content of the Pain Relief Kit with a member of the research staff. During this review the subject will be informed about the recommended use of all the four modes of the non-pharmacological interventions included in the kit. This information will also be included in written form in the Pain Relief Kit.
  Interventions: Behavioral: multimodal non-pharmacological Pain Relief Kit

INTERVENTIONS:
Behavioral: multimodal non-pharmacological Pain Relief Kit — Participants will be told: "No two people have the same kind of pain and that pain management must be individualized to your pain. Thus, we want you to try the four modes of the non-pharmacological interventions included in the kit individually and in combination in order to determine what works best to relieve your pain"
  The Pain Relief kit will also include written instructions and materials for three behavioral techniques directed at maintaining compliance with the non-pharmacological interventions. During the review of the Pain Relief Kit with a member of the research staff participants will be informed about the recommended use of the three behavioral techniques including setting goals, working with a buddy and keeping a graph of your progress. This information will also be included in written form in the Pain Relief Kit.

SUMMARY:
The purpose of this project is to determine the effect of a multimodal non-pharmacological Pain Relief Kit on the pain, functioning, patient satisfaction, and opioid consumption of individuals suffering from an acute pain episode of chronic neck and/or low back pain over a 3-week duration.

DETAILED DESCRIPTION:
The purpose of this project is to determine the effect of a multimodal non-pharmacological Pain Relief Kit on the pain, functioning, patient satisfaction, and opioid consumption of individuals suffering from an acute pain episode of chronic neck and/or low back pain over a 3-week duration. A secondary purpose of this study is to determine the effect of the kit on product sales and self-reported disability compared to patients who were not offered the kit.

Study Design: A convenience sample of 30 subjects who report being treated by a health care professional for musculoskeletal pain of an acute episode of chronic neck and/or low back pain which has lasted longer than 4 weeks will be recruited. Following screening for inclusion and exclusion criteria eligible individuals will provide informed consent prior to any data collection taking place. Following providing informed consent, subjects will engage in the baseline data collection protocol. Then after completing baseline data collection all participants will receive the intervention that includes the Pain Relief Kit for 3 weeks. All participants enrolled in the project will complete data collection at 3 data collection points. Baseline data collection will take place following informed consent. The second data collection point will take place one week following baseline data collection (T1) and the third data collection point will take place 3 weeks following baseline data collection (T2). In addition, all participants will provide a daily rating of their pain and documentation of pain management interventions they engaged in from the Pain Relief Kit, over the counter (OTC) treatments &/or treatments prescribed by a health care provider. This will result in a one group repeated measures design in which eligible participants will be provided with a Pain Relief Kit for 3 weeks.

Analysis: Repeated measures ANOVA will determine if the participants changed on any of the outcome variables over the duration of the project (p<.05). This analysis will be repeated to determine the impact of treatment compliance rates on the outcome variables. Main or interaction effects detected by the R-ANOVA will be explored further through calculated Tukey's post hoc comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18 and report experiencing average daily musculoskeletal pain of moderate intensity (>3/10) in the neck or low back for greater than 4 weeks.

Exclusion Criteria:

* Report any indication for medical clearance prior to engaging in moderate intensity exercise or if they have any other health limitations to engaging in moderate exercise.
* Additional exclusion criteria are the individual is unable to complete any of the data collection protocols, has previously been diagnosed with schizophrenia, dementia or is mentally incapable of providing informed consent or report a previous allergic reaction to kinesiotape or menthol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Medical Outcomes Study (MOS)-36 Physical functioning scale at 3 weeks | 3 (Baseline, 1 week, 3 weeks)
Change in visual analog scale (VAS) of pain at 3 weeks | 3 (Baseline, 1 week, 3 weeks)
Change in Timed performance of functional tasks at 3 weeks | 3 (Baseline, 1 week, 3 weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sport and Spine Rehab, Fairfax, Virginia
  - Sport and Spine Rehab, McLean, Virginia

IPD SHARING:
Plan to Share IPD: No